CLINICAL TRIAL: NCT04734002
Title: Neonatal Surgery Intensive Care Unit: Hacettepe Experience
Acronym: NSICUHE
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, H. Tolga Çelik, associate professor, Hacettepe University
Other Study IDs: GO-SURGERY
Record Dates: First submitted 2021-01-20; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Neonatal Surgery; Surgery--Complications; Newborn Morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Surgical treatment in the neonatal period mostly consists of congenital anomalies. Due to the different characteristics of newborns, the practice of monitoring this group of patients by neonatal specialists in neonatal intensive care units is increasingly common in the world and in our country. In our hospital, neonatal surgery intensive care unit model has been applied for about six years.

Objectives: This study was aimed at examining the data gathered from the neonatal surgery intensive care unit we created at Ihsan Dogramaci Children's Hospital and the contribution of this model toward improving the health of newborns with surgical problems.

Methods: The file records of newborns admitted to the neonatal and neonatal surgery intensive care units which operate on two separate floors at Ihsan Dogramaci Children's Hospital were retrospectively analyzed for the period January 2014 to December 2019. The information of the patients was recorded retrospectively for the study period with the information obtained from the hospital database.

The investigators believe that the neonatal surgery intensive care unit model should become widespread in Turkey. As there is a paucity of information concerning this subject in the literature worldwide and in our country, through this study the investigators wanted to draw attention to the subject by sharing our own experience working at İhsan Dogramaci Children's Hospital.

DETAILED DESCRIPTION:
Background: Surgical treatment in the neonatal period mostly consists of congenital anomalies. Due to the different characteristics of newborns, the practice of monitoring this group of patients by neonatal specialists in neonatal intensive care units is increasingly common in the world and in our country. In our hospital, neonatal surgery intensive care unit model has been applied for about six years.

Objectives: This study was aimed at examining the data gathered from the neonatal surgery intensive care unit we created at Ihsan Dogramaci Children's Hospital and the contribution of this model toward improving the health of newborns with surgical problems.

Methods: In this study, the file records of newborns admitted to the neonatal and neonatal surgery intensive care units which operate on two separate floors at Ihsan Dogramaci Children's Hospital were retrospectively analyzed for the period January 2014 to December 2019. The demographic, neonatal, and clinical information of the patients-including medical and surgical diseases and mortality rates-was recorded retrospectively for the study period with the information obtained from the hospital database. In addition, the gestational week, birth weight, gender, and length of hospital stay of the patients who were operated on in our unit in the last 2 years were examined.

The data obtained from the hospital database were recorded in Microsoft Excel and SPSS 22.0 Base, and statistical analysis was performed.

Aİm: This study was aimed at examining the data gathered from the neonatal surgery intensive care unit we created at Ihsan Dogramaci Children's Hospital and the contribution of this model toward improving the health of newborns with surgical problems.

ELIGIBILITY:
Inclusion Criteria:

* Newborns hospitalized in the Hacettepe University neonatal intensive care unit.
* All newborns who had surgery.

Exclusion Criteria:

* Babies older than 28 days.
* babies not recorded in the hospital database.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns hospitalized in the Hacettepe University neonatal intensive care unit. The file records of newborns admitted to the neonatal and neonatal surgery intensive care units which operate on two separate floors at Ihsan Dogramaci Children's Hospital were retrospectively analyzed for the period January 2014 to December 2019. The information of the patients was recorded retrospectively for the study period with the information obtained from the hospital database.
Sampling Method: Non-Probability Sample
Enrollment: 5442 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Neonatal Surgery Intensive Care Unit working principle | five years
  This study was aimed at examining the data gathered from the neonatal surgery intensive care unit the investigators created at Ihsan Dogramaci Children's Hospital and the contribution of this model toward improving the health of newborns with surgical problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddharth V, Gupta SK, Agarwala S, Satpathy S, Goel P. Outcome of Care Provided in Neonatal Surgery Intensive Care Unit of a Public Sector Tertiary Care Teaching Hospital of India. J Indian Assoc Pediatr Surg. 2019 Oct-Dec;24(4):257-263. doi: 10.4103/jiaps.JIAPS_177_18. PMID 31571756